CLINICAL TRIAL: NCT06099535
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Multicenter Study of LNK01001 Capsule in Moderately to Severely Active Rheumatoid Arthritis Patients With Inadequate Response or Intolerance to csDMARDs
Brief Title: A Study of LNK01001 Capsule in Moderately to Severely Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lynk Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LNK01001-2020-02RA
Record Dates: First submitted 2023-10-10; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LNK01001 Dose A (Experimental): Participants will receive LNK01001 Dose A orally BID for up to 24 weeks.
  Interventions: Drug: LNK01001 Dose A
- LNK01001 Dose B (Experimental): Participants will receive LNK01001 Dose B orally BID for up to 24 weeks.
  Interventions: Drug: LNK01001 Dose B
- placebo/LNK01001 Dose A (Placebo Comparator): Participants will receive a placebo orally BID for 12 weeks in Period 1. Participants will be re-randomized at Week 13 in a 1:1 ratio to receive LNK01001 Dose A orally BID for up to 24 weeks.
  Interventions: Drug: LNK01001 Dose A; Drug: placebo
- placebo/LNK01001 Dose B (Placebo Comparator): Participants will receive a placebo orally BID for 12 weeks in Period 1. Participants will be re-randomized at Week 13 in a 1:1 ratio to receive LNK01001 Dose B orally BID for up to 24 weeks.
  Interventions: Drug: LNK01001 Dose B; Drug: placebo

INTERVENTIONS:
Drug: LNK01001 Dose A — Capsules taken orally
  Arms: LNK01001 Dose A; placebo/LNK01001 Dose A
Drug: LNK01001 Dose B — Capsules taken orally
  Arms: LNK01001 Dose B; placebo/LNK01001 Dose B
Drug: placebo — Capsules taken orally
  Arms: placebo/LNK01001 Dose A; placebo/LNK01001 Dose B

SUMMARY:
This study includes two periods. In Period 1, Participants who meet eligibility criteria will be randomized in a 1:1:1 ratio to receive a twice-daily oral LNK01001 Dose A or LNK01001 Dose B or a matching placebo for 12 weeks. Participants who receive a placebo in Period 1 will be re-randomized at Week 13 in a 1:1 ratio to receive a twice-daily oral LNK01001 Dose A or LNK01001 Dose B for 12 weeks (period 2). Participants who receive LNK01001 ( Dose A and Dose B) in Period 1 will maintain the treatment dose in Period 2.

DETAILED DESCRIPTION:
This study includes a 35-day screening period; a 12-week randomized, double-blind, parallel-group, placebo-controlled treatment period (Period 1); a 12-week double-blind period (Period 2); and a 28 to 35-day follow-up period (FU).

Participants who meet eligibility criteria will be randomized in a ratio of 1：1：1 to 3 treatment groups in period 1， the placebo group will be rerandomized in a 1:1 ratio to LNK01001 Dose A or LNK01001 Dose B at week 13.

1. Group 1: LNK01001 Dose A BID (Day 1 to Week 12)， LNK01001 Dose A BID (Week 13 and thereafter)
2. Group 2：LNK01001 Dose B BID (Day 1 to Week 12)， LNK01001 Dose B BID (Week 13 and thereafter)
3. Group 3: Placebo (Day 1 to Week12) ， LNK01001 Dose A BID (Week 13 and thereafter)
4. Group 4: Placebo (Day 1 to Week12) ， LNK01001 Dose B BID (Week 13 and thereafter)

Participants who complete the Week 12 visit (end of Period 1) will enter Period 2, and continue to receive LNK01001 Dose A or Dose B treatment. Starting at Week 12, rescue therapy is allowed.

ELIGIBILITY:
Inclusion Criteria:

* Participants between ≥ 18 and ≤70 years of age.
* Diagnosis of RA for ≥ 3 months at screening visit who also fulfill the 2010 American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) classification criteria for RA.
* ≥ 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) at Screening and baseline visit.
* High-sensitivity C-Reactive Protein (hsCRP) ≥ ULN at Screening.
* Participants have been receiving csDMARD therapy ≥ 3 months and on a stable dose for ≥ 4 weeks prior to the first dose of study drug.

Exclusion Criteria:

* Subjects who are allergy to any component of the study drug.
* Subjects who are ACR functional class IV or long-term bedridden/long-term wheelchair.
* Prior exposure to Janus Kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
* Subjects who received intra-articular, intramuscular, intravenous, trigger point or tender point, intracapsular, or intra-tendon injections of glucocorticoids within 8 weeks before randomization.
* Current use of oral or inhaled glucocorticoids and the daily dose is >10 mg of prednisone (or equivalent dose) or on a not stable dose within 4 weeks before randomization.
* Current use of Non-steroidal anti-inflammatory drugs and on a not stable dose within 4 weeks before randomization.
* Subjects who received iguratimod treatment within 4 weeks before randomization.
* Subjects who received interferon treatment within 4 weeks before randomization.
* Current diagnosis of systemic inflammatory disease other than RA.
* History of malignancy or current diagnosis of malignancy within 5 years before screening visit.
* Uncontrolled diabetes, hypertension, kidney disease, liver disease, severe heart disease.
* Subject with any major surgery within 4 weeks before randomization or planned major surgery during study; history of chronic pain that may affect study evaluation; previous recipient of an organ transplant.
* Any clinically significant laboratory or ECG abnormal value, as determined by the Investigator, may interfere with the evaluation of the study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response at week 12 | week 12
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. 20% improvement in 68-tender joint count;
  2. 20% improvement in 66-swollen joint count; and
  20% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Health Assessment Questionnaire - Disability Index (HAQ-DI)
  * High-sensitivity C-reactive protein (hsCRP).

SECONDARY OUTCOMES:
Percentage of Participants With an ACR50 | Week1,2,4,8,12
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR50 response criteria:
  1.50% improvement in 68-tender joint count; 2.50% improvement in 66-swollen joint count; and 3.50% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Health Assessment Questionnaire - Disability Index (HAQ-DI)
  * High-sensitivity C-reactive protein (hsCRP).
Percentage of Participants With an ACR20 | Week1,2,4,8
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR20 response criteria:
  1. 20% improvement in 68-tender joint count;
  2. 20% improvement in 66-swollen joint count; and
  20% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Health Assessment Questionnaire - Disability Index (HAQ-DI)
  * High-sensitivity C-reactive protein (hsCRP)
Change From Baseline in Disease Activity Score 28 (DAS28)-CRP | Week1,2,4,8,12
  The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity
Change From Baseline in Disease Activity Score 28 (DAS28)-ESR | Week1,2,4,8,12
  The DAS28 is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and ESR. Scores on the DAS28 range from 0 to approximately 10, where higher scores indicate more disease activity
Change from Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI). | Week1,2,4,8,12
  The Health Assessment Questionnaire - Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. A negative change from Baseline in the overall score indicates improvement.
Percentage of Participants With an ACR70 | Week1,2,4,8,12
  Participants who met the following 3 conditions for improvement from baseline were classified as meeting the ACR70 response criteria:
  1. 70% improvement in 68-tender joint count; 2. 70% improvement in 66-swollen joint count; and 3.70% improvement in at least 3 of the 5 following parameters:
  * Physician global assessment of disease activity
  * Patient global assessment of disease activity
  * Patient assessment of pain
  * Health Assessment Questionnaire - Disability Index (HAQ-DI)
  * High-sensitivity C-reactive protein (hsCRP).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China